CLINICAL TRIAL: NCT04961749
Title: Retention of Whole-body Training Effects on Ambulatory Function in Children With Cerebral Palsy
Acronym: CP_WBVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Jeffrey Eggleston, Assistant Professor, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1745950-2
Record Dates: First submitted 2021-06-23; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: CP; Gait Disorders, Neurologic; Locomotion Disorder, Neurologic
Keywords: Cerebral Palsy; Locomotion; Pediatrics
MeSH Terms: conditions — Gait Disorders, Neurologic; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration group (Experimental): This group will receive vibration stimulation while standing on a side-alternating vibration platform. Vibration sessions will occur three times per week over four-weeks. Each session will include three-minutes of vibration followed by three-minutes rest, completing this sequence three times per session
  Interventions: Other: Whole body vibration training
- Control group (No Intervention): This group will not receive vibration, but will rather hear a recording of the vibration, while still standing on the vibration platform. Still, this group will receive this training three times per week over four-weeks with a similar three-minute rotation as the vibration group.

INTERVENTIONS:
Other: Whole body vibration training — Whole-body vibration training applies a vibration stimulus to an individual as they are standing on a side-alternating platform. The vibration creates small muscle contractions in the lower extremity musculature which has been shown to improve function and ambulatory function.
  Arms: Vibration group

SUMMARY:
This study will evaluate the retention effects of a four-week whole-body vibration training intervention in children with Cerebral Palsy. The primary outcomes for this study are gait function, including Timed Up and Go and the two-minute walk test. Secondary outcomes of this study include lower extremity gait function, coordination, and gait variability. For this study, a total of 10 children with Cerebral Palsy (CP) will be recruited with 5 being randomly placed into an experimental group and 5 being randomly placed into a control group. Each participant, regardless of group, will complete pre-, post-, and retention testing, with a four-week whole-body vibration training intervention between the pre- and post-testing. The four-week whole-body vibration training will include three visits per week, with the experimental group receiving a vibration stimulus while standing on a vibration platform. Vibration sessions will consist of three-minutes of vibration, followed by three minutes rest, completing this cycle three separate times. The control group will follow a similar pattern, but rather than experiencing vibration, they will hear a sound of the vibration platform through a speaker. Once the four-week training session is finished, participants will return after a three-month retention period to determine whether ambulation function was retained.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy
* Ability to walk independently

Exclusion Criteria:

* Musculoskeletal injuries or conditions (other than Cerebral Palsy) which alter their independent walking ability

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-06-16 (Estimated); Study Completion 2022-06-16 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test | 16 weeks
  Amount of time to quickly and safely complete the test
Two-minute walk test | 16 weeks
  Distance covered while walking for two minutes

SECONDARY OUTCOMES:
Lower extremity gait function | 16 weeks
  Three-dimensional motion capture will be used to track lower extremity segment movement patterns. All measurements will have units of degrees

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Eggleston, PhD, Principal Investigator — The University of Texas at El Paso
Locations (1):
- The University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT04961749/ICF_000.pdf